CLINICAL TRIAL: NCT03763279
Title: Suture of the Abdominal Wall With Triclosan-coated Polydioxanone Barbed Suture vs Triclosan-coated Polydioxanone Monofilament vs Polydioxanone Monofilament in Emergency Surgery
Brief Title: Effect of Barbed Suture and Triclosan-coated Monofilament in Emergency Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC-HUSJ 18-10
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the epidemiology nurse, who will assess the presence of SSI, will be blinded to the treatment assigned.
  The surgeon is masked to the assignment prior to consenting and enrolling the patient and initiating the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triclosan-coated barbed suture (Experimental): Abdominal wall closure will be performed using a Triclosan-coated Polydioxanone barbed suture
  Interventions: Combination Product: Triclosan-coated barbed suture
- Triclosan-coated monofilament suture (Experimental): Abdominal wall closure will be performed using a Triclosan-coated Polydioxanone monofilament suture
  Interventions: Combination Product: Triclosan-coated monofilament suture
- Monofilament suture (Sham Comparator): Abdominal wall closure will be performed using a monofilament suture
  Interventions: Device: Monofilament suture

INTERVENTIONS:
Combination Product: Triclosan-coated barbed suture — Use of Triclosan-coated Polydioxanone barbed suture
  Arms: Triclosan-coated barbed suture
Combination Product: Triclosan-coated monofilament suture — Use of Triclosan-coated Polydioxanone monofilament suture
  Arms: Triclosan-coated monofilament suture
Device: Monofilament suture — Use of Polydioxanone monofilament suture
  Arms: Monofilament suture

SUMMARY:
Patients will be randomized 3 groups:

Group 1: Abdominal fascial closure will be performed with Triclosan-coated barbed Polydioxanone suture

Group 2:Abdominal fascial closure will be performed with Triclosan-coated monofilament Polydioxanone suture

Group 3: Abdominal fascial closure will be performed with monofilament Polydioxanone suture

Incisional surgical.site infection and evisceration will be recorded.

DETAILED DESCRIPTION:
Patients will be randomized 3 groups:

Group 1: Abdominal fascial closure will be performed with Triclosan-coated barbed Polydioxanone suture (Stratafix Symmetric, J&J), caliber 1, 48mm-cylindric needle.

Group 2:Abdominal fascial closure will be performed with Triclosan-coated Polydioxanone loop suture (PDS plus looc, J&J), caliber 1, 48mm-cylindric needle.

Group 3: Abdominal fascial closure will be performed with Polydioxanone loop suture (PDS plus looc, J&J), caliber 1, 48mm-cylindric needle.

Incisional surgical.site infection and evisceration will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Contaminated and Dirty surgery
* Emergency surgery performed by midline laparotomic approach
* The following diagnosis will be included:

  * Anastomotic leak of previous digestive surgery (colon, small bowel or gastric surgery)
  * Colonic or bowel perforations
  * Appendicitis with purulent of fecal peritonitis, undergoing midline laparotomy
  * Perforation of gastric or duodenal ulcer
  * Intestinal ischemia requiring bowel resection

Exclusion Criteria:

* Emergency surgery undergoing laparoscopic approach
* Appendicitis operated by McBurney incision
* Intestinal isquemia without requiring bowel resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of incisional surgical-site infection | 30 days postoperatively
  Diagnosis of incisional surgical-site infection during the postoperative course

SECONDARY OUTCOMES:
Rate of Evisceration | 30 days postoperatively
  Diagnosis of evisceration during the postoperative course, which will be assessed by physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Andres Garcia-Marin, Study Director — Hospital de San Juan
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Llavero C, Jimenez-Fuertes M, Duran M, Perez-Lopez M, Garcia-Marin A. Incisional Surgical Site Infection after Abdominal Fascial Closure with Triclosan-Coated Barbed Suture vs Triclosan-Coated Polydioxanone Loop Suture vs Polydioxanone Loop Suture in Emergent Abdominal Surgery: A Randomized Clinical Trial. J Am Coll Surg. 2020 May;230(5):766-774. doi: 10.1016/j.jamcollsurg.2020.02.031. Epub 2020 Feb 27. PMID 32113031